CLINICAL TRIAL: NCT02619955
Title: Hepcicor Cohort : Clinical, Biological, Genetic and Fonctional charactérization of Rare Iron Overlaod phénotypes Associated With Hepcidin Deficiency Excluding C282Y Homozygosity
Brief Title: Cohort of Patients With Rare Iron Overloads Excluding C282Y Homozygosity
Acronym: HEPCICOR
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC14_9841
Record Dates: First submitted 2015-11-16; First posted 2015-12-02 (Estimated); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Rare Iron Overlaods
Keywords: hepcidin deficiency; genetic; except C282Y Homozygosity
MeSH Terms: interventions — DNA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Rare iron overload with hepcidin deficiency: clinical, biological, and genetic analysis of rare iron overlaod phenotype (except C282Yhomozygisity), samples with DNA
  Interventions: Other: samples with DNA

INTERVENTIONS:
Other: samples with DNA

SUMMARY:
The study explores the hepcidin deficiency causes of rare iron overload (excluding C282Y homozygosity), and aim to characterize this iron overload in term of clinical, biological, genetic and functional spacificities.

DETAILED DESCRIPTION:
Chronic iron overload are responsible for morbidity and mortality. There are many causes, genetic and acquired. Hepcidin deficiency related to genetic desease is one of them.

This study concerns specifically this cause, and seeks to characterize these iron overloads on clinical, biological, genetic and functional point of view.

A significant number of patients with chronic iron overload, present a phenotype of hepcidin deficiency. This profile is characterized by an elevated plasma iron increased serum transferrin saturation, a transferrin saturation, and a parenchyma distribution of iron overload. These diseases either remains unexplained or are associated with mutations in the gene involved in iron metablism regulation.

The main objective of this study is to characterize these iron overloads with phenotype of hepcidin deficiency not related to homozygosity C282Y (clinical, biological and genetic).

ELIGIBILITY:
Inclusion Criteria:

* Biological profile suggestive of hepcidin deficiency:

  * increase of transferrin saturation coefficient (> 50 %) verified on at least 2 times, and calculated from the transferrinemia.
  * Proved hepatic iron overload: by the dosage of the iron hepatic concentration either on block hepatic biopsic, or by MRI according to the method of quantification of the iron validated overload (by adopting a threshold of 100 µmol /g)
  * Patient's written consent for examination of genetic characteristics for diagnosis and collection development for genetic and not genetic research within the framework of an abnormality of the iron metabolism
  * Patient written inform consent.

Exclusion Criteria:

* HFE hemochromatosis: homozygosity C282Y/C282Y
* Treatment with iterative phlebotomy
* Hematologic diseases with dyserythropoiesis and/or repeated transfusions
* Haptoglobin low, below normal directing towards the diagnosis of chronic hemolysis, myelodysplasia
* Prolonged oral or parenteral iron supplementation
* Current or past excessive regular drinking
* Patient minor or under legal protection measure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting a rare iron overloads with hepcidin deficiency
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2023-01 (Actual); Study Completion 2023-01 (Actual)

PRIMARY OUTCOMES:
Number of patients presenting with mutation in gene know to be associated with iron metabolism | Inclusion
  to characterize these iron overloads with phenotype of hepcidin deficiency not related to homozygosity C282Y (clinical, biological and genetic).

SECONDARY OUTCOMES:
comparison of the hepcidin and hepcidin/ferritin ratio in patient with or without in gene known to be associated with iron metabolism | inclusion
  To Identificate potential explanatory factors of hepcidino deficiency phenotype
Number of patients presenting with associated causes of iron overload | inclusion
  - Identification of potentially explanatory factors visceral consequences of iron overload in hepcidino deficiency phenotype (overweight, high blood pressure, diabetes)
Genotype-Phenotype correlation | Inclusion
  To Research correlations genotype-phenotype
Hepatic and splenic iron concentration measurements by NMR | Inclusion
  Validation of the hepatic iron concentration measurements imaging ( nuclear magnetic resonance (NMR)) in the various centers
Number of patients with detectable abnormal iron species in blood (non transferrin bound iron, labile pool iron) | Inclusion
  - Assessment of the clinical value of biomarkers of iron metabolism

CONTACTS AND LOCATIONS:
Overall Officials: Edouard BARDOU-JACQUET, MD/PhD, Principal Investigator — CHU Pontchaillou
Locations (9):
- France (9):
  - CHU Limoges - Médecine interne A, Limoges
  - Centre Hospitalier Lyon-Sud, Lyon
  - CHRU de Montpellier - Hôpital St Eloi, Montpellier
  - Hôpital Hasenrain, Mulhouse
  - Hopital E.Muller, Mulhouse
  - CHR La Source, Orléans
  - Bardou Jacquet, Rennes
  - CHU Purpan, Toulouse
  - Hopital Paul Brousse, Villejuif